CLINICAL TRIAL: NCT04463485
Title: Impact of Umbilical Cord Clamping Time on Infant Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Sevil Güner, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Delayed Cord Clamping RCT
Record Dates: First submitted 2020-07-04; First posted 2020-07-09 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Third Stage of Labor; Healthy; Umbilical Cord Clamping Time; Infant Conditions
Keywords: umbilical cord; clamping; infant; anemia; midwifery
MeSH Terms: conditions — Anemia | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Clamping (Experimental): The intervention group was waited 60 seconds for umbilical cord clamping in the second stage of labor.
  Interventions: Procedure: Delayed Clamping
- Early Clamping (No Intervention): No interventions have been assigned.

INTERVENTIONS:
Procedure: Delayed Clamping — Umbilical cord clamping was delayed 60 seconds at the end of second stage of labor.
  Arms: Delayed Clamping

SUMMARY:
This research was conducted to carry out the effect of umbilical cord clamping time on baby anemia.

DETAILED DESCRIPTION:
This study is an experimental, randomized controlled study. The sample of the study consisted of 65 pregnant women and newborns (intervention=32, control=33) who applied for delivery at Ege University Medical Hospital Gynecology and Obstetrics Clinic at the time of the study. In this study, "Descriptive Data Form of Impact of Umbilical Cord Clamping Time on Infant Anemia" was used as a data collection tool. In the intervention group waited 60 seconds for umbilical cord clamping in the second stage of labor, in the control group the umbilical cord was clamped in the first 15 seconds. For the data of the first stage of the study, the neonatal hematocrit and bilirubin measurements and the need for phototherapy due to hyperbilirubinemia were evaluated 48 hours after birth. In the second stage of the study, data on anaemia screening performed in family medicine at the end of the fourth month of birth were examined. Statistical analysis of the data from the study was performed using IBM SPSS Statistics 25.0 package program. Parametric tests were used for statistical analysis of the data with a normal distribution. The level of statistical significance was determined as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Apply for normal birth
* Singleton pregnancy and live fetus
* Cephalic presentation
* Estimated birth weight between 2500-4000 grams
* Birth rates <5
* Women who received iron support during pregnancy
* Haemoglobin level ≥ 11 gr/dL
* No systemic disease or pregnancy complication that may pose a risk for postpartum bleeding.
* Neonates who don't need for resuscitation after birth
* Babies who did not receive iron supplements up to the 4th month after birth were included.

Exclusion Criteria:

* Pregnant women who refuse to participate in the research
* Neonates who need for resuscitation after birth
* Babies who receive iron supplements up to the 4th month after birth were excluded.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Neonatal Haematocrit Value at 48th Hours of Life | 48th hours after birth
  Haematocrit measurement in capillary blood taken from newborn after birth
Neonatal Bilirubin Value at 48th Hours of Life | 48th hours after birth
  Bilirubin measurement in capillary blood taken from newborn after birth
Phototherapy Requirement Rates due to Hyperbilirubinemia | 3 or 14 days of age
  Neonatal phototherapy requirement due to hyperbilirubinemia in the postpartum period
Haemoglobin Values of 4 Month Infants | Infants' 4th month of age
  Haemoglobin measurement at baby's 4th month of age
Haematocrit Values of 4 Month Infants | Infants' 4th month of age
  Haematocrit measurement at baby's 4th month of age
Diagnosis of Anemia Rates of 4 Month Infants | Infants' 4th month of age
  Screening of the family medicine center, condition of the baby diagnosed with anemia at 4th month of age

CONTACTS AND LOCATIONS:
Overall Officials: Birsen Saydam, Study Director — Ege University
Locations (1):
- Ege University Medical Hospital Obstetric and Gynecology Department, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.